CLINICAL TRIAL: NCT00428350
Title: A 24-Week, Multi-Centre, Open-Label, Single-Arm, Phase IV Study of the Efficacy and Safety of Seroquel (Quetiapine Fumarate) With Daily Dose 600mg-750mg as Mono-Therapy in the Treatment of Acute Schizophrenic Patients
Brief Title: Study of Efficacy and Safety of Seroquel (Quetiapine Fumarate) as Mono-Therapy for Acute Schizophrenic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00004; SOLO
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine Fumarate (Seroquel)

SUMMARY:
The primary objective of the study is to evaluate the efficacy of quetiapine fumarate (Seroquel) with daily dose 600mg-750mg used as mono-therapy in the treatment of acute schizophrenic patients by evaluation of the change from baseline in PANSS total score at Day 56 using the last observation carried forward (LOCF) method.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent for study participation before initiation of any study related procedures, signed by the patient's legal guardian
* Female and/or male, aged between 18 and 60 years (inclusive)
* Is hospitalised in a psychiatric unit with an acute episode of schizophrenia defined by CCMD-3 criteria as one of the following: [20.1] paranoid schizophrenia, [20.2] hebephrenic schizophrenia, [20.3] catatonic schizophrenia, [20.5] undifferentiated schizophrenia

Exclusion Criteria:

* CCMD-3 diagnosis of mental retardation
* Psychosis judged to be the direct physiological effect of an abused medication or substance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-12; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in PANSS total score at Day 56 (LOCF)

SECONDARY OUTCOMES:
Change from baseline in PANSS positive scale score at Day 56 (LOCF)
Change from baseline in PANSS negative scale score at Day 56 (LOCF)
Change from baseline in PANSS EC score at day 56 ,
Change from baseline in MADRS total score at Day 56. etc

CONTACTS AND LOCATIONS:
Overall Officials: Jon Zhu, MD, Study Director — AstraZeneca; Gang Wang, MD, Principal Investigator — Beijing An Ding hospital
Locations (9):
- China (9):
  - Research Site, Guangzhou, Guangdong
  - Research Site, Harbin, Heilongjiang
  - Research SIte, Wuhan, Hubei
  - Research Site, Nanjing, Jiangsu
  - Research Site, Jinan, Shandong
  - Research Site, Kunming, Yunnan
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Huzhou, Zhejiang
  - Research Site, Beijing